CLINICAL TRIAL: NCT00060970
Title: Restoration of Muscle Function During Rehabilitation
Brief Title: Evaluating Muscle Function After Ankle Surgery
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: R29HD033738 (NIH)
Record Dates: First submitted 2003-05-16; First posted 2003-05-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Muscle Atrophy; Muscle Weakness; Fractures
Keywords: Disuse atrophy; Ankle fracture; Exercise, therapy; Cast immobilization; Deconditioning; Sarcopenia
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness; Fractures, Bone; Muscular Disorders, Atrophic; Ankle Fractures; Motor Activity; Sarcopenia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Physical Therapy

SUMMARY:
Patients who are forced to rest or reduce activity as a result of illness, injury, or surgery often experience resulting muscle weakness. This study will evaluate muscle features and muscle strength in patients who are recovering from surgery for broken ankles. The goal of this study is to improve the recovery of muscle function and overall ability after prolonged periods of ankle inactivity due to surgery.

DETAILED DESCRIPTION:
Many physiological conditions are associated with muscle weakness and can affect movement. This study will investigate which metabolic and morphological features of skeletal muscle are uniquely altered during the course of rehabilitation and how they affect muscle function and performance in daily ambulatory activities. This study will also examine how well the commonly used assessment measures reflect actual muscle capacity. Finally, because there is evidence that activity does not affect all fiber types uniformly, fiber-type specific metabolic and morphological measures will be performed.

Participants in this study will have had an ankle injury that has been treated surgically (Open Reduction Internal Fixation, or ORIF) followed by 5 to 10 weeks of cast immobilization. Following initial baseline measurements made after 1 week of re-ambulation, participants are enrolled in a 10-week rehabilitation program that focuses on restoration of both muscle strength and endurance. Assessments are made at Weeks 5 and 10 and include 31P-Magnetic Resonance Spectroscopy (MRS), Magnetic Resonance Imaging (MRI), muscle biopsy, and muscle function and functional performance tests. 31P-measurements monitor changes in the in vivo metabolic characteristics of skeletal muscle. 3D-MRI procedures will be used to quantify the maximal muscle cross-sectional area and total muscle volume. Muscle endurance and strength will be measured using an isokinetic dynamometer. Functional performance tests consist of self-selected walking pace, power for ascending and descending stairs, and toe raises while standing on one foot.

Nine participants (six patients and three control volunteers) will be studied each year. Control volunteers are submitted to the same measurements at similar time intervals in order to assess variability over time.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 10 weeks of cast immobilization following surgery (ORIF) for mallerolar fracture

Exclusion Criteria:

* Pregnant or breastfeeding
* Severe claustrophobia
* MRI incompatible metal implants (e.g., pacemaker)
* Diabetes or peripheral neuropathies
* Bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1995-09; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Krista Vandenborne, Ph.D., P.T., Principal Investigator — University of Pennsylvania, Department of Physiology
Locations (1):
- MMRRCC, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Elliott MA, Walter GA, Gulish H, Sadi AS, Lawson DD, Jaffe W, Insko EK, Leigh JS, Vandenborne K. Volumetric measurement of human calf muscle from magnetic resonance imaging. MAGMA. 1997 Jun;5(2):93-8. doi: 10.1007/BF02592238. PMID 9268071
- [Background] Vandenborne K, Elliott MA, Walter GA, Abdus S, Okereke E, Shaffer M, Tahernia D, Esterhai JL. Longitudinal study of skeletal muscle adaptations during immobilization and rehabilitation. Muscle Nerve. 1998 Aug;21(8):1006-12. doi: 10.1002/(sici)1097-4598(199808)21:83.0.co;2-c. PMID 9655118
- [Background] Elliott MA, Walter GA, Swift A, Vandenborne K, Schotland JC, Leigh JS. Spectral quantitation by principal component analysis using complex singular value decomposition. Magn Reson Med. 1999 Mar;41(3):450-5. doi: 10.1002/(sici)1522-2594(199903)41:33.0.co;2-9. PMID 10204865
- [Background] Shaffer MA, Okereke E, Esterhai JL Jr, Elliott MA, Walker GA, Yim SH, Vandenborne K. Effects of immobilization on plantar-flexion torque, fatigue resistance, and functional ability following an ankle fracture. Phys Ther. 2000 Aug;80(8):769-80. PMID 10911415
- [Background] Gregory CM, Vandenborne K, Dudley GA. Metabolic enzymes and phenotypic expression among human locomotor muscles. Muscle Nerve. 2001 Mar;24(3):387-93. doi: 10.1002/1097-4598(200103)24:33.0.co;2-m. PMID 11353424
- See also: Click here for more information about the Metabolic Magnetic Resonance Research and Computing Center, University of Pennsylvania — http://www.siuh.edu